CLINICAL TRIAL: NCT00335192
Title: Determination of Plasma and Intracellular Levels of Nucleoside Reverse Transcriptase Inhibitors (NRTI) and of Nucleotide Analog Tenofovir Disoproxil Fumarate (TDF) in Patients Treated With Abacavir and/or Lamivudine Given With or Without TDF.
Brief Title: To Determine if There Are Pharmacokinetic Interactions at Plasma or Intracellular Level Between Nucleosides and Tenofovir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: LLuita Sida Foundation, LLuita Sida Foundation
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INTRANUCS; 2004-000948-25
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: HIV
Keywords: Intracellular concentrations; Plasma concentration; Abacavir; Tenofovir; Lamivudine (3TC); Pharmacokinetic interactions
MeSH Terms: interventions — Therapeutics; Lamivudine; lopinavir-ritonavir drug combination; VBA protocol; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Phase I: 3TC + TDF + NVP or LPV/rtv
  Phase II: patients on treatment with LPV/rtv, stop TDF during 4 weeks: 3TC + LPV/rtv
  Interventions: Drug: Patients in treatment with 3TC + TDF + LPV/rtv, stop tenofovir during 4 weeks
- 2 (Experimental): Phase I: ABV + TDF + NVP or LPV/rtv
  Phase II: patients on treatment with LPV/rtv, stop TDF during 4 weeks: ABV + LPV/rtv
  Interventions: Drug: Patients in treatment with ABV + TDF + LPV/rtv, stop tenofovir during 4 weeks
- 3 (Experimental): Phase I: 3TC + ABV + TDF + NVP or LPV/rtv
  Phase II: patients on treatment with LPV/rtv, stop TDF during 4 weeks: 3TC + ABV + LPV/rtv
  Interventions: Drug: Patients in treatment with 3TC + ABV + TDF+ LPV/rtv, stop TDF during 4 weeks

INTERVENTIONS:
Drug: Patients in treatment with 3TC + TDF + LPV/rtv, stop tenofovir during 4 weeks — 3TC (300 mg/24 h, 1 tablet/24 h) + Lopinavir/ritonavir (400 mg/12 h, 3 tablets/12 h)
  Other Names: Epivir; Kaletra
  Arms: 1
Drug: Patients in treatment with ABV + TDF + LPV/rtv, stop tenofovir during 4 weeks — ABV (300 mg/12 h, 1 tablet/12 h)+ Lopinavir/ritonavir (400 mg/12 h, 3 tablets/12 h)
  Other Names: Ziagen; Kaletra
  Arms: 2
Drug: Patients in treatment with 3TC + ABV + TDF+ LPV/rtv, stop TDF during 4 weeks — 3TC (300 mg/24 h, 1 tablet/24 h)+ ABV (300 mg/12 h, 1 tablet/12 h)+ Lopinavir/ritonavir (400 mg/12 h, 3 tablets/12 h).
  Other Names: Epivir; Ziagen; Kaletra
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate if there are pharmacokinetic interactions between the NRTI 3TC and ABV, and the TDF nucleotide. For this purpose, the intracellular and plasma levels of 3TC and ABV will be compared in patients given these nucleosides with TDF and 30 days after the interruption of the TDF.

DETAILED DESCRIPTION:
There is clear evidence of pharmacokinetic interaction between ddI+TDF. However, the interaction between TDF and other NRTIs, mainly at intracellular level, has not been so well studied.

Since all the NRTIs are anabolized at intracellular level by numerous kinases, and are transported by passive carrier systems, the interaction may be between TDF and other NRTIs.

This study aims to investigate the pharmacokinetic interactions between the TDF and the nucleosides abacavir (ABV) and lamivudine (3TC) at plasma and intracellular level.

With this objective, intracellular and plasma levels will be analysed in a group of patients that receive the combinations 3TC +TDF, ABV+TDF and 3TC+ABV+TDF together with lopinavir/rtv or nevirapine. Subsequently, in a second phase of the study, in the group of patients given ABV and/or 3TC + TDF + lopinavir/rtv, the pharmacokinetic determinations will be repeated after a 4-week interruption of the TDF .

ELIGIBILITY:
Inclusion Criteria:

1. HIV+ patients aged above 18 years.
2. Undetectable HIV viral load in the last determination
3. Patients capable of correct compliance according to clinical criteria.
4. Patients on triple HAART therapy for the previous 3 months including 3TC and/or ABV and TDF, with a PI (Lopinavir/ritonavir) or an NNRTI (Nevirapine)
5. Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use a barrier contraceptive method during the study.
6. Ability to provide informed consent.

Exclusion Criteria:

1. Incorrect therapeutic compliance over the four weeks before the beginning of the study.
2. Interruption or withdrawal from therapy during follow-up.
3. Concomitant treatment with any drug which according to the clinician's criterion may interact with the investigational antiretrovirals, such as other antiretrovirals.
4. Triple HAART therapy including Nevirapine (for phase II)
5. Documented or suspected resistance to ABV, 3TC or lopinavir/rtv (for phase II).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the variation between the intracellular levels of 3TC and ABC before and after the interruption of the treatment with TDF | At baseline and week 4.

SECONDARY OUTCOMES:
Variations between the plasma levels of 3TC and ABC before and after interruption of the treatment with TDF. | at baseline and week 4
Correlation between the intracellular and plasma levels of 3TC, ABC and TDF. | at baseline and week 4
Changes in the intracellular levels of TDF following the withdrawal of the drug. | At week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unit
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain